CLINICAL TRIAL: NCT02551120
Title: Characterization of Patients With Idiopathic Hypoparathyroidism, Autosomal Dominant Hypocalcaemia and Pseudohypoparathyroidism
Brief Title: Characterization of Patients With Non-surgical Hypoparathyroidism and Pseudohypoparathyroidism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Lars Rejnmark, Professor, DMSci, PhD, University of Aarhus
Other Study IDs: M-20110074-2
Record Dates: First submitted 2015-06-17; First posted 2015-09-16 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Idiopathic Hypoparathyroidism; Autosomal Dominant Hypocalcaemia; Pseudohypoparathyroidism
Keywords: Idiopathic hypoparathyroidism; Autosomal dominant hypocalcaemia; Pseudohypoparathyroidism; Quality of Life; Bone Mineral Density; Muscle strength; Cardiovascular indices
MeSH Terms: conditions — Hypoparathyroidism; Hypercalciuric Hypocalcemia, Familial; Pseudohypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (whole blood, serum and plasma), urine collection (24h) and bone biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with idiopathic hypoparathyroidism, autosomal dominant hypocalcaemia and pseudohypoparathyroidism.

SUMMARY:
Hypoparathyroidism (hypoPT) and pseudohypoparathyroidism (Ps-hypoPT) are rare diseases, characterized by low levels of parathyroid hormone [PTH] and plasma calcium or high plasma PTH and low plasma calcium, respectively. A recently study by the investigators' group, identified 123 living persons with idiopathic hypoPT and 62 living persons with Ps-hypoPT, only few of these have been genetic tested.

The aim of the study is to perform a detailed clinical and genetic characterization of Danish patients with idiopathic hypoPT and Ps-hypoPT. Patients will be examined by questionnaires, biochemistry, scans, bone biopsies and genetic tests. Furthermore the investigators aim to perform family tracing for the hereditary forms. The prevalence of magnesium depletion will be assessed as well.

In addition to providing new information on symptoms, co-morbidity, and prognosis for this group of patients, the investigators presume that the study may improve their understanding on calcium homeostasis and bone metabolism in general.

DETAILED DESCRIPTION:
Background:

Hypoparathyroidism (HypoPT) is a group of rare clinical disorders characterized by hypocalcaemia and hyperphosphatemia with inappropriate low levels of parathyroid hormone (PTH). Due to the lack of PTH, the renal production of 1α,25-dihydroxycholecalciferol (1,25(OH)2D) is reduced. Most often, HypoPT is caused by accidental removal of the parathyroid glands during neck surgery (postsurgical hypoPT). However, in rare in-stances HypoPT is caused by autoimmune disorders with immune mediated destruction of the parathyroid glands, or a variety of genetic mutations, including the CATCH-22 (DiGeorge) Syndrome, familial isolated HypoPT or an activating mutation in the gene encoding the calcium-sensing receptor (CaSR), termed autosomal dominant hypocalcaemia (ADH).

The CaSR is not only found in the parathyroid glands, but is also expressed by other tissue including the renal tubules. Low plasma levels of ionised calcium (Ca2+) are registered by the calcium sensing receptors (CaSR) located e.g. in the cell membranes of the parathyroids and in the renal tubules. Low levels of Ca2+ increases the release of PTH from the parathyroids, which normalises plasma Ca2+ and decrease P-phosphate. Lack of PTH decreases the renal synthesis of 1,25-dihydroxycholecalciferol, witch in combination with low PTH decreases bone turnover. Although, large-scale meta-analysis of genome wide association data incorporating 150 candidate genes did not link the CaSR to bone mineral density or osteoporotic fracture risk, no specific data are available on whether BMD in patients with an activating mutation in their CaSR gene (ADH patients) differs from the general population. The largest case series of patients with ADH so far reported included 25 patients and did not report BMD within this group.

Calcium is of importance to many physiological processes, including cardiovascular functioning. The CaSR has been suggested to be of importance in the regulation of blood pressure and a Batter's like phenotype has been reported in patients with ADH. Although the recent study by the investigators' group did not show an increased cardiovascular morbidity in patients with postsurgical hypoPT, no data are available on blood pressure regulation or indices of atherosclerosis in patients with idiopathic hypoPT.

PseudoHypoPT is due to PTH resistance in the target organs, causing hypocalcemia with inappropriate high PTH concentrations. The phenotype in type 1 is known as Albrights's hereditary osteodystrophy, (AOH) (maternal 2 of 8 allele). Pseudo-pseudoHypoPT is characterized by AOH, but without the typical biochemical findings (pater-nal allele). PseudoHypoPT type 2 has typical biochemical changes but no characteristic phenotype. Discrepant results have been reported on effects on bone mineral density (BMD), as some studies has shown a decreased BMD (hyperparathyroid bone disease), whereas other studies have shown that BMD actually may be increased.

Untreated, hypoPT is characterized by an increased neuromuscular irritability including weakness, muscle cramps, paraesthesias of the lips, tongue, fingers and feet, loss of memory, headaches and uncontrollable cramping muscle movements of the wrists and feet (carpopedal spasm). Other symptoms may be spasm of the facial muscles (Chovstek´s Sign) and the contraction of the muscle produced by ischemia (Trousseaus Sign).

In long standing congenital cases there may be cataract and malformations of the teeth's. Due to high blood phosphorous levels intracranial calcifications (basal ganglia) may be seen by X-ray. Renal stones and renal failure may develop either because of the disease or its treatment. Studies have shown that postsurgical hy-poPT is associated with a reduced quality of life (QoL).

Aim:

The aim of the project is to perform a detailed clinical and genetic characterization of Danish patients with idiopathic hypoparathyroidism, including pseudohypoparathyroidism. Patients will be examined as detailed in the section on methods, and genetic tests will be performed in patients who have not been tested previously. Furthermore the investigators aim to perform family tracing for the hereditary forms.

Design:

A cross-sectional descriptive study on patients with idiopathic hypoparathyroidism, autosomal dominant hypocalcaemia and pseudohypoparathyroidism, including family tracing for inherited forms.

Materials and methods:

Study subjects:

All patients with non-surgical hypoPT in Denmark will be invited by letter to participate in the study. Patients who accept participation will undergo a detailed examination in terms of:

* Questionnaire/ interviews:
* Quality of life: To study the participants health related quality of life the WHO's 5 Well-Being Index, the Physical Activity Scale (PAS), and the SF-36v2 will be used in a Danish version.
* Biochemistry incl. genetics
* 24hours urine:
* Cardiovascular indices: Blood pressure is measured in sitting position twice after minimum 5 minutes of rest. The presence of atherosclerosis is assessed by tonometry measuring pulse wave velocity and central aortic pressure using the SphygmoCor System.
* Muscle function- and postural stability: Isometric maximum voluntary muscle strength on the dominant hand side is measured using a dynamometer connected to a computer (Good Strength TM, Meititur Ldt, Finland) (25;26). Muscle strength is assessed at knee and elbow flexion and extension. Similarly, grip strength on the dominant hand is measured. Balance function is assessed by measuring the dynamic stability on a stadiometer (Meititur Ltd, Finland). Two smaller physical tests are also performed, "Repeated chair stand test" and "Timed Up and Go-test".
* Osteodensitometry: Bone mineral content (BMC) and areal bone mineral density (aBMD) is assessed by Dual-Energy X-ray absorptiometry" (DXA) using a Hologic Discovery scanner. Measurements are performed at the lumbar spine (L1-L4), hip region, forearm, and the whole body. Furthermore, body composition (lean and fat-tissue mass) will be determined by DXA. Volumetric total, cortical, and trabecular bone mineral density (vBMD) at the lumbar spine (L1+L2) and at the hip are assessed using quantitative computer tomography (QCT) (Mid-ways Software Inc., Austin Texas, USA). Bone microarchitecture is assessed by high resolution peripheral quantitative computer tomography (HRpQCT)-scans of the right forearm and tibia using an XtremeCT scanner (Scan-co Medical).
* Bone biopsies: a bone biopsy will be obtained from the iliac crest for histomorphometric analyses. Prior to the biopsy, intravital tetracycline double marking will be performed.
* Family tracing: Investigations on first degree relatives will be performed in patients with known inherited forms of hypoPT as well as in patients with hypoPT of unknown origin. At first, family members will have plasma levels of calcium and PTH measured. If results show signs of hypoPT, the relatives will be examined as the index persons themselves (as detailed in this protocol).

Statistics:

Differences between study groups are assessed using Fisher's Exact Test for categorical variables and a two-sample t-test or Mann-Whitney U-test for continuous variables, as appropriate. Sample size calculation are as detailed in the section on hypothesis.

Ethical considerations:

The general protocol has been approved by the Central Denmark Region Committees on Biomedical Research Ethics.

Perspective:

HypoPT is a rare disease and only few data are available on this group of patients. In addition to providing new information on symptoms, co-morbidity, and prognosis for this group of patients, the investigators presume that the study may improve their understanding on mechanisms of importance to calcium homeostasis and bone metabolism in general.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either:

Idiopathic hypoparathyroidism, pseudohypoparathyroidism or autosomal dominant hypocalcaemia

* Participants must be able to read and understand Danish

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with non-surgical hypoPT and pseudohypoparathyroidism in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-08 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Study of patients (clinical characterization) with idiopathic hypoPT, ADH and pseudohypoPT | 3 years
  A detailed clinical characterization of Danish patients with idiopathic HypoPT, ADH and Ps-HypoPT including genetics of patients with idiopathic HypoPT and Ps-HypoPT.

SECONDARY OUTCOMES:
Quality of Life (QoL) | 3 years
  SF-36 version 2
Quality of Life (QoL) | 3 years
  WHO-5 Well Being Index
Bone Mineral Density (BMD) | 3 years

OTHER OUTCOMES:
Postural stability | 3 years
Blood pressure | 3 years
  Blood pressure, measured three times after 10 min rest.
Arterial stiffness as measured by tonometry | Three years
  Indices of arterial stiffness
Genetic characterization | Three years
  Patients with no known mutation, are offered a genetic screening for the most common mutations known.
Muscle strength and balance as measured by isometric tests and dynamic stability tests | Three years
  Effects on muscle strength (isometric tests of flexion and extension of thigh and hand), two function-tests (timed up-and go and timed stand-and-sit), and postural stability

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, DmSci, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided